CLINICAL TRIAL: NCT03862079
Title: Randomized Phase II Trial of Total Gut Decontamination Followed by Fecal Microbiota Transplant (FMT), FMT-Alone or Standard of Care for Reduction in Acute Graft-Versus-Host Disease of the Gastrointestinal Tract in Patients Given Broad-Spectrum Antibiotics
Brief Title: Fecal Transplant +/- Gut Decontamination in Preventing Acute Graft Versus Host Disease in Patients Given Broad-Spectrum Antibiotics
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Per PI's request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-0466; NCI-2019-01045 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0466 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Graft-versus-host Disease Prevention
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Fecal Microbiota Transplantation; Nystatin; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (TGD + FMT) (Experimental): Patients receive piperacillin-tazobactam PO TID and nystatin QID. Patients undergo stem cell transplantation on day 0, then undergo FMT via enema over 5-10 minutes within 3 weeks after transplantation.
  Interventions: Procedure: Fecal Microbiota Transplantation; Drug: Nystatin; Drug: Piperacillin-Tazobactam
- Arm II (FMT) (Experimental): Patients undergo stem cell transplantation on day 0, then undergo FMT via enema over 5-10 minutes within 3 weeks after transplantation.
  Interventions: Procedure: Fecal Microbiota Transplantation
- Arm III (standard therapy) (Active Comparator): Patients receive standard of care.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: Best Practice — Given standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm III (standard therapy)
Procedure: Fecal Microbiota Transplantation — Undergo FMT
  Other Names: Fecal Material Transplantation; Fecal Transplantation; FMT; Poo Transplant; Poop Transplant; Stool Transplant
  Arms: Arm I (TGD + FMT); Arm II (FMT)
Drug: Nystatin — Given PO
  Other Names: Mycostatin; Nystex
  Arms: Arm I (TGD + FMT)
Drug: Piperacillin-Tazobactam — Given PO
  Other Names: PIPER/TAZO; Piperacillin/Tazobactam; Zosyn
  Arms: Arm I (TGD + FMT)

SUMMARY:
This phase II trial studies how well a fecal microbiota transplant with or without total gut decontamination works in preventing graft versus host disease in patients exposed to broad-spectrum antibiotics. Fecal microbiota transplantation is the administration by enema of fecal matter (stool) that includes helpful bacteria from a normal, healthy donor. Total gut decontamination uses antibiotics to remove/reduce the amount of bacteria in the digestive system. It is not yet known if a fecal microbiota transplant with or without total gut decontamination works better in preventing graft versus host disease compared to standard immunosuppressive therapies (therapies that lower the normal function of the immune system).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients who develop acute graft-versus-host disease (GVHD) of the gastrointestinal (GI) tract by day 100 post-transplant for patients randomized to the standard of care, total gut decontamination (TGD) followed by fecal microbiota transplant (fecal microbiota transplantation [FMT]) and FMT alone arms.

SECONDARY OBJECTIVES:

I. Overall maximum stage of lower GI tract GVHD by day 100 post-transplant. II. Cumulative incidence of acute GVHD grade II-IV and maximum grade through 6 months.

III. Time to onset of acute GVHD and acute GI GVHD. IV. Incidence of adverse events and serious adverse events. V. Incidence of bacterial blood stream infections through 6 months. VI. Hematologic recovery (neutrophils and platelets). VII. Characterization of the intestinal microbiota at enrollment, pre-FMT / time of engraftment, 2 month post-FMT/ engraftment, onset of gastrointestinal tract (GIT) GVHD, and at study completion (6 months).

VIII. Relapse-free survival at 6 months post-randomization. IX. Non-relapse mortality at 6 months post-randomization. X. Overall survival (OS) at 6 months post-randomization.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM A (TGD + FMT): Patients receive piperacillin-tazobactam orally (PO) three times daily (TID) and nystatin PO four times daily (QID) until FMT. Patients undergo stem cell transplantation on day 0, then undergo FMT via enema over 5-10 minutes within 3 weeks after transplantation.

ARM B (FMT): Patients undergo stem cell transplantation on day 0, then undergo FMT via enema over 5-10 minutes within 3 weeks after transplantation.

ARM C (STANDARD THERAPY): Patients receive standard of care.

After completion of study treatment, patients are followed up at 100 days and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are day -10 pre- to day +30 post-allogeneic hematopoietic cell transplant (AHCT) from any donor or graft source and for any conditioning regimen
* Patients who have received treatment with meropenem or piperacillin-tazobactam (pip-tazo) intravenously (IV) (of at least 24 hours duration) in past 7 days
* Controlled infection defined as hemodynamically stable and not requiring supplemental oxygen of more than 2 liters via nasal cannula
* Patients who are able to take oral medications in suspension form
* Patients who are able to provide informed consent (IC) and comply with all study visits and procedures

Exclusion Criteria:

* Patients who are anticipated to require continued broad spectrum antibiotics with meropenem or pip-tazo IV for > 96 hours post-engraftment such as for known, documented infections necessitating prolonged treatment
* Patients with a prior documented infection with mycormycetes
* Patients who are greater than 2 days from time of neutrophil engraftment post AHCT
* Patients with active enteric infections
* Patients with acute GVHD >= grade II
* Patients unwilling or unable to undergo the FMT via retention enema procedure
* Patients who have received treatment with an investigational agent within 2 weeks of enrollment
* Patients unable to tolerate oral decontamination regimen of pip-tazo and nystatin due to prior allergy or intolerance of these medications
* Patients with any medical or psychological condition that, in the opinion of the investigator, might interfere with the subject's participation in the trial, pose any additional risk for the subject, or confound the assessments of the subject

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of acute gastrointestinal (GI) graft versus host disease (GVHD) | Within 100 days from time of transplant
  Summary statistics, including mean, median, range, and standard deviation, will be provided for continuous variables. Frequency tables will be used to summarize categorical variables.
Relapse-free survival | At 6 months post-randomization
  Relapse is defined by either morphological or cytogenetic evidence of acute leukemia or myelodysplastic syndrome (MDS) inconstant with pre-transplant features, or radiologic evidence of lymphoma, documented or not by biopsy. The distribution of time-to-event endpoints, as well as the median and 90% confidence interval, will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Microbiome diversity | At 2 weeks post fecal microbiota transplantation (FMT) (or engraftment for control arm)
  Will be measured using the inverse Simpson index. Summary statistics, including mean, median, range, and standard deviation, will be provided for continuous variables. Frequency tables will be used to summarize categorical variables.
Overall maximum stage of lower GI tract GVHD | Within 100 days post-transplant
  Will be defined as the proportion of patients who do not develop GI GVHD within 100 days post-transplant and will be monitored simultaneously in cohorts of 5 patients separately in each arm using the approach of Thall, Simon, and Estey.
Cumulative incidence of acute GVHD grade II-IV and maximum grade | Up to 6 months
  Summary statistics, including mean, median, range, and standard deviation, will be provided for continuous variables. Frequency tables will be used to summarize categorical variables.
Incidence of adverse and serious adverse events | Within 60 days of FMT
  Defined as the proportion of patients who develop blood stream infections caused by enteric bacteria within 60 days of FMT. Will be monitored simultaneously in cohorts of 5 patients separately in each arm using the approach of Thall, Simon, and Estey.
Incidence of bacterial blood stream infections | Up to 6 months
  Will identify those caused by a potential enteric pathogen. Summary statistics, including mean, median, range, and standard deviation, will be provided for continuous variables. Frequency tables will be used to summarize categorical variables.
Hematologic recovery (neutrophils and platelets) | Up to 6 months
  Summary statistics, including mean, median, range, and standard deviation, will be provided for continuous variables. Frequency tables will be used to summarize categorical variables.
Characterization of the intestinal microbiota | Baseline up to 6 months
  Summary statistics, including mean, median, range, and standard deviation, will be provided for continuous variables. Frequency tables will be used to summarize categorical variables.
Non-relapse mortality | At 6 months post-randomization
  Relapse is defined by either morphological or cytogenetic evidence of acute leukemia or MDS inconstant with pre-transplant features, or radiologic evidence of lymphoma, documented or not by biopsy. The distribution of time-to-event endpoints, as well as the median and 90% confidence interval, will be estimated using the Kaplan-Meier method.
Overall survival | At 6 months post-randomization
  The distribution of time-to-event endpoints, as well as the median and 90% confidence interval, will be estimated using the Kaplan-Meier method.

OTHER OUTCOMES:
Analysis of T-cell subsets | Up to 6 months post-enrollment
  Analysis of T-cell subsets (including specifically regulatory T-cells) will be performed by characterization of peripheral blood flow cytometry.
Analysis of serum/stool butyrate levels | Up to 6 months post-enrollment
Assessment of gut permeability | At time of discontinuation of antibiotics (engraftment)
  Will be performed via lactulose/ mannitol assay.

CONTACTS AND LOCATIONS:
Overall Officials: Amin M Alousi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org